CLINICAL TRIAL: NCT06213584
Title: The Effectiveness of Mulligan and Proprioceptive Neuromuscular Fasciliation Techiniques in Rotator Cuff Pathology: A Randomized Controlled Double-blind Study.
Brief Title: Mulligan and Proprioceptive Neuromuscular Fasciliation Techiniques in Rotator Cuff Pathology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Gamze Aydin, Istanbul Okan University, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IOU
Record Dates: First submitted 2024-01-10; First posted 2024-01-19 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Rotator Cuff Injuries
Keywords: rotator cuff injuries; mulligan mobilization; proprioceptive neuromuscular fascilitation; pain; functionality; quality of life
MeSH Terms: conditions — Rotator Cuff Injuries; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- mulligan mobilization (Experimental): Mulligan mobilization techniques
  Interventions: Other: conservative rehabilitation; Other: mullgan mobilization techniques
- pnf (Experimental): Proprioceptive neuromuscular fasciliation techniques
  Interventions: Other: conservative rehabilitation; Other: pnf
- conservative rehabilitation (Experimental): Conservative rehabilitation
  Interventions: Other: conservative rehabilitation

INTERVENTIONS:
Other: conservative rehabilitation — Hotpack + TENS + streching exercises
Other: mullgan mobilization techniques — Passive mobilization techniques during active movements
  Arms: mulligan mobilization
Other: pnf — hold relax active movements
  Arms: pnf

SUMMARY:
The aim of this study is to investigate the effects of Mulligan Mobilization techniques, Mobilization with Movement (MWMs) and Proprioceptive Neuromuscular Facilitation (PNF) techniques, Hold-Relax Active Movement Technique, on pain, normal joint range of motion, proprioception, scapular dyskinesia and functional status in individuals with rotator cuff syndrome.

A total of 60 people were included in the study: 20 participants in the censervative rehabilitation group (Conservative Treatment), 20 participants in the Treatment A (Mulligan Mobilization Application) Group, and 20 participants in the Treatment B (PNF Application) Group. Individuals were treated for 5 days for 4 weeks. Pain before and after treatment with Visual Analog Scale; joint range of motion with goniometer; With proprioception Angle Repetition Test; Scapular dyskinesia with Lateral Scapular Slide Test; quality of life with SF-36; shoulder functionality was assessed with the Western Ontario Rotator Cuff Scale (WORC).

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 25-75,
* diagnosed with rotator cuff syndrome,
* patients who did not have any obstacle to the evaluation parameters

Exclusion Criteria:

* having had shoulder surgery,
* presence of scoliosis,
* presence of cardiac pacemaker,
* history of recent myocardial infarction,
* presence of malignancy,
* corticosteroid treatment within the last 3 months

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-01-05 (Actual); Primary Completion 2021-03-05 (Actual); Study Completion 2022-03-25 (Actual)

PRIMARY OUTCOMES:
goniometer | 12 months
  shoulder range of motion
visual analog scale | 12 months
  shoulder pain intensity
angle repetition test | 12 months
  proprioception
lateral scapular glide test | 12 months
  presence of scapular dyskinesia
Western Ontario Rotator Cuff Index | 12 months
  functionality
SF-36 | 12 months
  quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Gamze AYDIN, Principal Investigator — Okan University
Locations (1):
- Istanbul Okan University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No